CLINICAL TRIAL: NCT07371611
Title: Sintilimab Plus Chemotherapy as Neoadjuvant and Adjuvant Treatment for Locally Advanced Oral Squamous Cell Carcinoma: A Multicenter, Open-label, Randomized, Phase III Clinical Study
Brief Title: Sintilimab Plus Chemotherapy as Neoadjuvant and Adjuvant Treatment for Locally Advanced Oral Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qunxing Li,MD (Other)
Responsible Party: Sponsor-Investigator, Qunxing Li,MD, Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-966-01
Record Dates: First submitted 2025-12-26; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Oral Squamous Cell Carcinoma; Oral Squamous Cell Carcinoma (OSCC)
Keywords: Oral Squamous Cell Carcinoma; Locally Advanced; Sintilimab; Perioperative Immunotherapy; Neoadjuvant Therapy; Adjuvant Therapy; Randomized Phase III Trial
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — sintilimab; 130-nm albumin-bound paclitaxel; Platinum Compounds; Carboplatin; Cisplatin; Radiotherapy; Chemoradiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Masking Description: This is an open-label study. No masking is applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Neoadjuvant sintilimab combined with TP regimen followed by radical surgery and risk-stratified adjuvant therapy (low-risk: sintilimab monotherapy; high-risk: radiotherapy or concurrent chemoradiotherapy followed by sequential sintilimab).
  Interventions: Drug: Sintilimab plus nab-paclitaxel and platinum-based chemotherapy
- Control arm (Active Comparator): Radical surgery combined with radiotherapy or chemoradiotherapy
  Interventions: Procedure: Radical surgery combined with radiotherapy or chemoradiotherapy

INTERVENTIONS:
Drug: Sintilimab plus nab-paclitaxel and platinum-based chemotherapy — Neoadjuvant sintilimab combined with TP regimen followed by radical surgery and risk-stratified adjuvant therapy (low-risk: sintilimab monotherapy; high-risk: radiotherapy or concurrent chemoradiotherapy followed by sequential sintilimab).
  Other Names: Sintilimab; Nab-paclitaxel; Carboplatin; Cisplatin
  Arms: Experimental arm
Procedure: Radical surgery combined with radiotherapy or chemoradiotherapy — Participants undergo radical surgical resection as primary treatment, followed by postoperative radiotherapy or concurrent chemoradiotherapy according to pathological risk factors and standard clinical practice.
  Other Names: surgery; radiotherapy; chemoradiotherapy
  Arms: Control arm

SUMMARY:
This is a multicenter, open-label, randomized phase III clinical trial evaluating perioperative treatment with sintilimab combined with chemotherapy in patients with locally advanced oral squamous cell carcinoma.

Despite standard treatment with surgery followed by postoperative radiotherapy or chemoradiotherapy, patients with locally advanced oral squamous cell carcinoma remain at high risk of recurrence or metastasis. Recent evidence, including results from the KEYNOTE-689 study, suggests that perioperative immunotherapy may improve survival outcomes, and this approach has been incorporated into NCCN guidelines. Combining immunotherapy with chemotherapy may further improve prognosis in this patient population.

Eligible participants will be randomly assigned to either an experimental group or a control group. The experimental group will receive neoadjuvant sintilimab combined with chemotherapy followed by surgery and postoperative treatment based on pathological response. Patients with major pathological response (MPR) will receive adjuvant sintilimab, while patients without MPR will receive postoperative radiotherapy or concurrent chemoradiotherapy combined with sintilimab. The control group will receive standard treatment consisting of surgery followed by postoperative radiotherapy or chemoradiotherapy as clinically indicated.

The primary objective of the study is to compare event-free survival between the two groups. Secondary objectives include overall survival, pathological response, safety, and treatment-related adverse events. The results of this study may help optimize perioperative treatment strategies and improve outcomes for patients with locally advanced oral squamous cell carcinoma.

DETAILED DESCRIPTION:
Oral squamous cell carcinoma (OSCC) is one of the most common malignancies of the head and neck region. A substantial proportion of patients present with locally advanced disease at diagnosis and remain at high risk of recurrence or metastasis despite radical surgery followed by postoperative radiotherapy or concurrent chemoradiotherapy. Previous studies have shown that conventional neoadjuvant or adjuvant chemotherapy provides limited benefit in improving long-term survival outcomes. Recent advances in immunotherapy have demonstrated significant efficacy in recurrent or metastatic head and neck squamous cell carcinoma, and emerging evidence supports the role of perioperative immunotherapy in resectable disease.

The KEYNOTE-689 study demonstrated that perioperative immunotherapy could improve event-free survival in patients with locally advanced, resectable head and neck squamous cell carcinoma, leading to the incorporation of this strategy into the National Comprehensive Cancer Network (NCCN) guidelines. However, further optimization of perioperative treatment strategies is required to enhance pathological response and survival outcomes, particularly in patients with locally advanced OSCC.

This study is a multicenter, open-label, randomized phase III clinical trial designed to evaluate the efficacy and safety of perioperative sintilimab combined with chemotherapy compared with standard treatment (surgery with or without postoperative radiotherapy or chemoradiotherapy) in patients with locally advanced OSCC. Eligible patients will be randomized in a 1:1 ratio to either the experimental group or the control group.

Patients in the experimental group will receive neoadjuvant sintilimab combined with chemotherapy prior to definitive surgical resection. Postoperative treatment will be stratified according to pathological response. Patients achieving major pathological response (MPR) will receive adjuvant sintilimab for at least six cycles or until unacceptable toxicity. Patients without MPR will receive postoperative radiotherapy or concurrent chemoradiotherapy sequentially combined with sintilimab for at least six cycles or until unacceptable toxicity. Patients in the control group will receive standard treatment consisting of surgical resection followed by postoperative radiotherapy or concurrent chemoradiotherapy as clinically indicated.

The primary endpoint of the study is event-free survival. Secondary endpoints include overall survival, pathological response to treatment, safety, and treatment-related adverse events. This study is expected to provide high-level evidence to optimize perioperative treatment strategies and improve clinical outcomes for patients with locally advanced oral squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years at the time of enrollment.
* ECOG Performance Status (PS) score of 0-1.
* Primary lesion pathologically confirmed as oral squamous cell carcinoma (OSCC), including tumors of the anterior two-thirds of the tongue, gingiva, buccal mucosa, floor of the mouth, hard palate, or retromolar trigone.
* Clinical stage III or IVA, defined as T1-2 with N1-2, or T3-4a and/or N0-2, according to the AJCC 8th edition OSCC TNM staging system.
* Willingness to undergo surgical treatment.
* Presence of at least one measurable lesion as defined by RECIST v1.1 criteria.
* Voluntary participation with full understanding and signing of the informed consent form, and willingness to comply with study procedures.
* Adequate major organ function, meeting all of the following laboratory criteria:
* 1. Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L without granulocyte colony-stimulating factor (G-CSF) administration within 14 days prior to testing.
* 2. Platelet count ≥ 100 × 10⁹/L without blood transfusion within the previous 14 days.
* 3. Hemoglobin > 90 g/L without blood transfusion or erythropoietin use within the previous 14 days.
* 4. Total bilirubin ≤ 1.5 × the upper limit of normal (ULN); ≤ 3 × ULN in cases of Gilbert's syndrome or non-hepatic indirect bilirubin elevation.
* 5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; ≤ 5 × ULN for patients with hepatic involvement.
* 6. Serum creatinine ≤ 1.5 × ULN and creatinine clearance (calculated by the Cockcroft-Gault formula) ≥ 60 mL/min.
* 7. Adequate coagulation function, defined as INR or prothrombin time (PT) ≤ 1.5 × ULN.
* 8. Normal thyroid function, defined as thyroid-stimulating hormone (TSH) within the normal range. Subjects with abnormal TSH may be enrolled if total T3 (or FT3) and FT4 are within normal limits.
* 9. Normal myocardial enzyme profile (minor laboratory abnormalities deemed clinically insignificant by the investigator are acceptable).
* 10. For women of childbearing potential, a negative urine or serum pregnancy test within 3 days prior to the first dose of study treatment (Cycle 1, Day 1) is required. If the urine test is indeterminate, a serum test must be performed. Non-childbearing women are defined as those who have been postmenopausal for at least one year or have undergone surgical sterilization or hysterectomy.
* 11. All participants (male or female) with reproductive potential must agree to use highly effective contraception (annual failure rate <1%) during the entire treatment period and for at least 120 days after the last study drug dose or 180 days after the last chemotherapy dose.

Exclusion Criteria:

* Prior treatment targeting PD-1, PD-L1, PD-L2, or CTLA-4, or other therapies targeting T-cell costimulatory or immune checkpoint pathways.
* Participation in another interventional clinical trial or use of an investigational drug or device within 4 weeks prior to the first dose.
* History of radiotherapy involving the head, neck, or maxillofacial regions.
* Use of traditional Chinese medicines or immunomodulatory agents with OSCC indications (e.g., thymosin, interferon, interleukin) within 2 weeks before first dosing; local therapy for pleural effusion control is permitted.
* History of active autoimmune disease within the past 2 years requiring systemic therapy (e.g., corticosteroids or immunosuppressants). Exceptions include:
* 1. Hypothyroidism controlled with thyroid hormone replacement therapy.
* 2. Diabetes mellitus controlled with insulin.
* 3. Adrenal or pituitary insufficiency treated with physiologic doses of corticosteroids.
* Use of immunosuppressive agents:
* 1. Systemic corticosteroid therapy within 1 week prior to the first dose is prohibited.
* 2. Use of other immunosuppressive drugs is prohibited.
* 3. Intranasal, inhaled, or topical corticosteroids are permitted.
* 4. Physiologic doses of corticosteroids (e.g., prednisone ≤10 mg/day or equivalent) are permitted.
* Prior systemic antitumor therapy, except patients who have had ≥12 months of treatment-free interval between the last chemotherapy and initiation of neoadjuvant therapy.
* Previous allogeneic organ or hematopoietic stem cell transplantation (excluding corneal transplantation).
* Known hypersensitivity to sintilimab, carboplatin, cisplatin, nab-paclitaxel, or any of their excipients.
* Failure to recover to baseline or ≤ grade 1 (except fatigue or alopecia) from adverse events or complications of prior interventions before enrollment.
* Known human immunodeficiency virus (HIV) infection (HIV-1/2 antibody positive).
* Untreated active hepatitis B infection (HBsAg positive with HBV-DNA above the ULN). Subjects meeting the following criteria may be enrolled:
* 1. HBV viral load <1000 copies/mL (200 IU/mL) and receiving antiviral therapy during the study to prevent reactivation.
* 2. Subjects who are anti-HBc(+), HBsAg(-), anti-HBs(-), and HBV-DNA(-) do not require prophylactic antiviral therapy but must be closely monitored for viral reactivation.
* Active hepatitis C infection (HCV antibody positive with HCV-RNA above the lower limit of detection).
* Receipt of a live vaccine within 30 days prior to the first dose (inactivated vaccines, such as inactivated influenza vaccine, are permitted; intranasal live vaccines are not allowed).
* Pregnant or breastfeeding women.
* Presence of severe or uncontrolled systemic diseases, including but not limited to:
* 1. Cardiac disorders: severe arrhythmias (e.g., complete left bundle branch block, second-degree or higher atrioventricular block, ventricular arrhythmia, or persistent atrial fibrillation), unstable angina, or congestive heart failure (NYHA class ≥ II).
* 2. Vascular disorders: history of unstable angina, myocardial infarction, transient ischemic attack, or stroke within 6 months before enrollment.
* 3. Poorly controlled hypertension (systolic BP >140 mmHg or diastolic BP >90 mmHg).
* 4. Pulmonary disorders: noninfectious pneumonitis requiring corticosteroid therapy within 1 year prior to the first dose, or active interstitial lung disease.
* 5. Infectious diseases: active infections requiring systemic treatment, or severe uncontrolled infections.
* 6. Active pulmonary tuberculosis.
* 7. Gastrointestinal disorders: clinically active diverticulitis, intra-abdominal abscess, or intestinal obstruction.
* 8. Hepatic disorders: liver cirrhosis, decompensated liver disease, or acute/chronic active hepatitis.
* 9. Poorly controlled diabetes mellitus: fasting blood glucose (FBG) >10 mmol/L.
* 10. Renal dysfunction: urine protein ≥++ on urinalysis and 24-hour urinary protein >1.0 g.
* 11. Psychiatric disorders: severe mental illness that may affect treatment compliance.
* Any other condition that, in the opinion of the investigator, makes the subject unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | 2 years
  Event-free survival is defined as the time from randomization to the first occurrence of disease progression, local or distant recurrence, second primary malignancy, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
overall survival（OS） | 2 years and 5 years.
  Overall survival (OS) was defined as the time from randomization to death from any cause.
pathological complete response（pCR） | At the time of definitive surgery
  Pathological complete response (pCR) is defined as the absence of residual viable tumor cells on microscopic examination in the resected primary tumor and lymph nodes, with all evaluated lymph nodes being negative. The pCR rate is calculated as the proportion of participants achieving pCR among all enrolled participants. The pCR rate is expressed as a percentage and its 95% confidence interval is estimated using the exact binomial distribution.
Major Pathological Response (MPR) | At the time of definitive surgery
  Major pathological response (MPR) is defined as the presence of 10% or less residual viable tumor cells in the resected primary tumor specimen on microscopic examination after neoadjuvant treatment, regardless of lymph node status. The MPR rate is calculated as the proportion of participants achieving MPR among all enrolled participants. The MPR rate is expressed as a percentage and its 95% confidence interval is estimated using the exact binomial distribution.
Treatment-related adverse events（TRAE） | through study completion, an average of 1 year
  Treatment-related adverse events (TRAEs) are defined as adverse events that are considered by the investigator to be possibly, probably, or definitely related to the study treatment, including sintilimab, chemotherapy, surgery, radiotherapy, or chemoradiotherapy. Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 6.0. The incidence, severity, and type of TRAEs will be summarized and analyzed.
Radiologic assessments | Baseline and preoperative
  Radiologic assessments are performed to evaluate tumor response using contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI). Tumor response is assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1, based on independent radiologic review.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Li, MD, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made publicly available. De-identified and aggregated data may be shared upon reasonable request to the corresponding author following publication, subject to approval and data use agreements.

REFERENCES:
- [Result] Uppaluri R, Haddad RI, Tao Y, Le Tourneau C, Lee NY, Westra W, Chernock R, Tahara M, Harrington KJ, Klochikhin AL, Brana I, Vasconcelos Alves G, Hughes BGM, Oliva M, Pinto Figueiredo Lima I, Ueda T, Rutkowski T, Schroeder U, Mauz PS, Fuereder T, Laban S, Oridate N, Popovtzer A, Mach N, Korobko Y, Costa DA, Hooda-Nehra A, Rodriguez CP, Bell RB, Manschot C, Benjamin K, Gumuscu B, Adkins D; KEYNOTE-689 Investigators. Neoadjuvant and Adjuvant Pembrolizumab in Locally Advanced Head and Neck Cancer. N Engl J Med. 2025 Jul 3;393(1):37-50. doi: 10.1056/NEJMoa2415434. Epub 2025 Jun 18. PMID 40532178